CLINICAL TRIAL: NCT05438693
Title: Factors Affecting Time Elapsed From First Symptom Till Complete Diagnosis of Multiple Sclerosis, Initiation of Disease Modifying Treatment and Drug Adherence in Upper Egypt
Brief Title: Delayed Diagnosis of Multiple Sclerosis, Treatment Initiation and Non-adherence in Upper Egypt
Status: Completed | Type: Observational
Sponsor: doaa mokhtar mahmoud (Other)
Responsible Party: Sponsor-Investigator, doaa mokhtar mahmoud, lecturer, Assiut University
Organization: Assiut University (Other)
Other Study IDs: SVU MED NAP020 2 20 7 56
Record Dates: First submitted 2022-06-16; First posted 2022-06-30 (Actual); Last update posted 2022-06-30 (Actual); Status verified 2022-06

CONDITIONS: Multiple Sclerosis, Relapsing-Remitting
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The earlier that MS can be diagnosed; the sooner treatment can be initiated with timely reduction of subclinical disease activity and prevention of disability progression.

However, significant delays can still occur between noticing the first symptoms and receiving a diagnosis even before a person with symptoms suggestive of MS sees a neurologist. Such delays could be due to heterogeneity of clinical and imaging manifestations, which not only differ between patients, but also vary in individual patients over time. Moreover, lack of awareness of the primary care physicians about MS presentations, the limited accessibility to specialized centers or the non-availability of diagnostic tools such as MRI scanners and lumbar puncture, may further add to this delay and increases the risk of disability.

There are also many factors that can contribute to delayed initiation of DMT after diagnosis like inadequate knowledge with DMT, their high coast and limited access to health care insurance services.

Like many chronic conditions, non- Adherence to drug therapies is estimated up to 50%, with associated increased morbidity, mortality, and health care costs.

To the best of our knowledge, this is the first study in upper Egypt that tries to address these factors. By conducting this study, we aim at identifying factors leading to delayed diagnosis of MS, initiation and adherence to DMT in order to translate recent advances in the diagnosis and treatment of MS into improved outcomes in the lives of people with MS and their families and to avoid many of the long-term economic and personal costs that result from unnecessary irreversible disability.

DETAILED DESCRIPTION:
this is cross-sectional study in the Neuropsychiatry department, South Valley university hospitals, where patients with remitting relapsing multiple sclerosis according to McDonald criteria 2017 using disease modifying treatment for at least 3 months are recruited. patients were recruited from 3 major MS clinics in Assiut, South valley and Luxor.

each patient was subjected to the following:

* Full history and neurological examination including EDSS scores.
* MRI brain and spine.
* Electrophysiologic study: VEP, ABR, SSEP.
* clinical scales:

  1. The Arabic version of the eight-item Morisky Medication Adherence Scale (MMAS-8).
  2. Treatment Satisfaction Questionnaire for Medication (TSQM-9).
  3. Extended disability status scale (EDSS) measurement for MS patients
  4. Hamilton depression rating-17-item version (HAM-D 17).
  5. Fatigue Severity Scale (FSS) for determination of fatigue degree using the Arabic validated version
  6. The Pittsburgh Sleep Quality Index (PSQI)
  7. International Restless Legs Syndrome rating scale time to diagnosis and DMT initiation was calculated and the rate of adherence was determined this was followed be determining factors related to each Data analysis was done using the IBM Statistical Package for Social Sciences software package version 20.0. (Armonk, NY: IBM Corp). The qualitative variables were described with ratio and percentage. The Shapiro-Wilk test was used to verify the normality of distribution. Quantitative variables with normal distribution were reported with mean and SD, and those without normal distribution were described using median and range of mid-quartiles. The level of statistical significance was set at p < 0.05.

The used tests were

1. - Chi-square test: For categorical variables, to compare between different groups
2. - Monte Carlo correction: Correction for chi-square when more than 20% of the cells have expected count less than 5
3. - Mann Whitney test: For abnormally distributed quantitative variables, to compare between two studied categories
4. - Kruskal-Wallis test: For abnormally distributed quantitative variables, to compare between more than two studied categories
5. - Regression: univariate and multivariate logistic regression for factors related to delayed diagnosis, delayed treatment initiation and non-adherence

ELIGIBILITY:
Inclusion Criteria:

* Patient with confirmed diagnosis of remitting relapsing multiple sclerosis according to the 2017 McDonald's criteria and receiving any DMT for at least 3 months.

Exclusion Criteria:

* Presence of any clinical or radiological finding suggesting a diagnosis other than MS or other demyelinating diseases.
* Presence of other systemic disease or being on long term treatment for any disease.
* Incomplete clinical or radiological data were provided.
* Subject declined to provide written informed consent.

Ages: 18 Years to 60 Years | Sex: All
Age Groups: Adult
Study Population: Eighty patients diagnosed with remitting relapsing MS and on DMTs were included in the study. MS was diagnosed based on the clinical examination, magnetic resonance imaging (MRI), lumbar puncture (LP), and visual evoked potential (VEP) using McDonald criteria. They were included according to the previous inclusion and exclusion criteria.
  all cases were interviewed and examined by a neurologist and the following data were retrospectively collected: demographic, clinical data, therapeutic history, complete clinical examination including EDSS score, radiological data, electrophysiological tests results and clinical scales including: MMAS-8, TSQM-9, PSQI, IRLS and FSS
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
time to diagnosis of multiple sclerosis | From date of first documented MS symptom until the date of first documented diagnosis, assessed up to 10 years from onset symptoms
  time to MS diagnosis is measured from the date of the first symptom till the date of the official diagnosis of MS
time to disease modifying treatment initiation | From date of first documented diagnosis until the date of first documented date of start of DMT, assessed up to 10 years from diagnosis
  time to DMT initiation is calculated from the date of diagnosis till the date the patient first received the prescribed DMT
rate of adherence to disease modifying treatment among MS patients | in the last month period prior to interview
  the rate of adherence to DMT among MS patients is measured by Morinski medical adherence scale for medications. with a score of 8 is considered adherent while <8 is considered non-adherent.

SECONDARY OUTCOMES:
determine factors related to delayed diagnosis of MS | From date of first documented MS symptom until the date of first documented diagnosis, assessed up to 10 years from onset symptoms
  after reviewing literature, a number of factors related to delayed diagnosis of MS were determined including (age, sex, residence, education, marital status, first presenting symptom, year of presentation , first medical specialty sought and previous misdiagnosis).
  the frequency of those risk factors in patients with both early and delayed diagnosis were calculated and bivariate and multivariable analysis indicated the possible independent predictive factors to the diagnostic delay
frequency of depression as a factor related to DMT adherence | in the last month period prior to interview
  the frequency of depression (using Hamilton depression scale-21), is measured and correlated to adherence. The score range from 0-50, Higher scores on this scale (>=8) are indicative of depression.
frequency of fatigue as a factor related to DMT adherence | in the last month period prior to interview
  the frequency of fatigue (using the fatigue severity scale-9), is measured and correlated to adherence. the score range from 1-63, Higher scores on this scale (>=36) are indicative of fatigue
frequency of sleep disturbances as a factor related to DMT adherence | in the last month period prior to interview
  the frequency of sleep disturbances (using Pittsburgh Sleep Quality Index), is measured and correlated to adherence. It consists of 19 self- rated questionnaires and 5 additional questionnaires for bed partner. It provides a global score of sleep on a scale from 1 to 21, with higher scores indicating more sleep complaints.
treatment satisfaction as a factor related to DMT adherence | in the last month period prior to interview
  treatment satisfaction (using Treatment Satisfaction Questionnaire for Medication-9), is measured and correlated to adherence. Questions comprise four aspects representing the personal impressions of treatment benefit, tolerability, convenience of use, and general satisfaction with the treatment. scores for each of the TSQM subscales ranged from 0 to 100. total Scores obtained were summed and the percentage of satisfaction score was calculated, where higher scores indicated higher satisfaction

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - South valley University, Qina, Qena Governorate
  - Assiut University, Asyut

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Koch-Henriksen N, Sorensen PS. The changing demographic pattern of multiple sclerosis epidemiology. Lancet Neurol. 2010 May;9(5):520-32. doi: 10.1016/S1474-4422(10)70064-8. PMID 20398859
- [Background] Giovannoni G, Butzkueven H, Dhib-Jalbut S, Hobart J, Kobelt G, Pepper G, Sormani MP, Thalheim C, Traboulsee A, Vollmer T. Brain health: time matters in multiple sclerosis. Mult Scler Relat Disord. 2016 Sep;9 Suppl 1:S5-S48. doi: 10.1016/j.msard.2016.07.003. Epub 2016 Jul 7. PMID 27640924
- [Background] Gaitan MI, Correale J. Multiple Sclerosis Misdiagnosis: A Persistent Problem to Solve. Front Neurol. 2019 May 7;10:466. doi: 10.3389/fneur.2019.00466. eCollection 2019. No abstract available. PMID 31133970
- [Background] Kaufmann M, Kuhle J, Puhan MA, Kamm CP, Chan A, Salmen A, Kesselring J, Calabrese P, Gobbi C, Pot C, Steinemann N, Rodgers S, von Wyl V; Swiss Multiple Sclerosis Registry (SMSR). Factors associated with time from first-symptoms to diagnosis and treatment initiation of Multiple Sclerosis in Switzerland. Mult Scler J Exp Transl Clin. 2018 Dec 6;4(4):2055217318814562. doi: 10.1177/2055217318814562. eCollection 2018 Oct-Dec. PMID 30559972
- [Background] McNicholas N, Hutchinson M, McGuigan C, Chataway J. 2017 McDonald diagnostic criteria: A review of the evidence. Mult Scler Relat Disord. 2018 Aug;24:48-54. doi: 10.1016/j.msard.2018.05.011. Epub 2018 Jun 21. PMID 29936325
- [Background] Ashur ST, Shamsuddin K, Shah SA, Bosseri S, Morisky DE. Reliability and known-group validity of the Arabic version of the 8-item Morisky Medication Adherence Scale among type 2 diabetes mellitus patients. East Mediterr Health J. 2015 Dec 13;21(10):722-8. doi: 10.26719/2015.21.10.722. PMID 26750162
- [Background] Vermersch P, Hobart J, Dive-Pouletty C, Bozzi S, Hass S, Coyle PK. Measuring treatment satisfaction in MS: Is the Treatment Satisfaction Questionnaire for Medication fit for purpose? Mult Scler. 2017 Apr;23(4):604-613. doi: 10.1177/1352458516657441. Epub 2016 Jul 11. PMID 27364322
- [Background] Hamilton M. Development of a rating scale for primary depressive illness. Br J Soc Clin Psychol. 1967 Dec;6(4):278-96. doi: 10.1111/j.2044-8260.1967.tb00530.x. No abstract available. PMID 6080235
- [Background] Al-Sobayel HI, Al-Hugail HA, AlSaif RM, Albawardi NM, Alnahdi AH, Daif AM, Al-Arfaj HF. Validation of an Arabic version of Fatigue Severity Scale. Saudi Med J. 2016 Jan;37(1):73-8. doi: 10.15537/smj.2016.1.13055. PMID 26739978
- [Background] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771
- [Background] Shalash AS, Elrassas HH, Monzem MM, Salem HH, Abdel Moneim A, Moustafa RR. Restless legs syndrome in Egyptian medical students using a validated Arabic version of the Restless Legs Syndrome Rating Scale. Sleep Med. 2015 Dec;16(12):1528-31. doi: 10.1016/j.sleep.2015.07.032. Epub 2015 Sep 25. PMID 26611951